CLINICAL TRIAL: NCT03222804
Title: Establishing a Milk Oriented Microbiota in Healthy Term Infants
Brief Title: Milk Oriented Microbiota
Acronym: MOM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not receive funding to start the trial.
Sponsor: University of California, Davis (Other)
Collaborators: Evolve BioSystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 738191
Record Dates: First submitted 2017-07-07; First posted 2017-07-19 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Microbial Colonization
Keywords: Infants; Probiotic; B. Infantis
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: The feeding patterns of eighty eligible infants (8 to 12 weeks in age) will be characterized based on a 7-day diet record that will be filled out by their mothers during the 7-day lead-in period starting with Day -7 and ending with Day -1. Of the eighty infants, twenty will be exclusive breast feeders (BF), twenty will be exclusive formula feeders (FF) and forty will be mixed-feeders (MF). Infants in all three feeding groups will consume B. infantis for twenty-one consecutive days. Participants will then enter the observational phase until their infant turns 1 year old.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exclusively breastfed (Active Comparator): Exclusive breastfeeding will be defined at screening as infants who have not consumed any infant formula after 7 days postnatal and have been exclusively breastfed without formula between day 7 of life through the end on the Lead-in period. ). Infants will consume B. infantis for twenty-one consecutive days.
  Interventions: Dietary Supplement: Bifidobacterium
- Exclusively formula fed (Active Comparator): Exclusive formula feeding is defined at screening as infants who consume only infant formula between day 7 of life through the end on the Lead-in period. Infants will consume B. infantis for twenty-one consecutive days.
  Interventions: Dietary Supplement: Bifidobacterium
- Mixed fed (Active Comparator): Mixed feeding is defined at screening as infants who consume a combination of infant formula and breast milk between day 7 of life through the end on the Lead-in period. Infants will consume B. infantis for twenty-one consecutive days.
  Interventions: Dietary Supplement: Bifidobacterium

INTERVENTIONS:
Dietary Supplement: Bifidobacterium — Each B. infantis (strain: BIEVC001) dose will be provided in one 625 mg sachet delivering 156 mg of live bacteria at a dose of 9x10^9 CFU plus 469 mg of pharmaceutical-grade lactose as the excipient and dispensed to participants by the study personnel.
  Other Names: B. infantis

SUMMARY:
The purpose of this study is to determine if supplementing healthy term infants delivered vaginally who consume breast milk, formula, or both with a probiotic for 21 consecutive days increases levels of bacteria in infants' stool.

DETAILED DESCRIPTION:
The purpose of phase 1 of this two phase clinical trial is to determine: 1) the effect of decreasing levels of human milk oligosaccharides on fecal B.infantis during and after 21 days of supplementation with Evolve activated B.infantis using exclusively breastfed, mixed-fed and exclusively formula-fed infants; 2) determine the effect of Evolve activated B.infantis on fecal B.infantis levels in exclusively breastfed infants compared to pre-supplementation levels.

ELIGIBILITY:
Inclusion Criteria:

* Women with infants age 8 to 12 weeks
* Term infants born >37 weeks gestation
* Mother-infant pairs who live within a 20-mile radius from UC Davis campus in Davis, CA or within a 20-mile UCDMC
* Women and infants who live in one location
* Infants born vaginally
* Infants who are either exclusively formula-fed, exclusively breastfed or mixed-fed
* Women who are mixed and formula feeding their infants who are willing to switch infant formulas and use the study's infant formula (Earth's Best Organic Infant Formula With Iron, Earth's Best) throughout the first two months of the study
* Women who are breastfeeding but introduce infant formula to their infants during the first two months of the study who are willing to use the study's infant formula (Earth's Best Organic Infant Formula With Iron, Earth's Best) for the first two months of the study

Exclusion Criteria:

* Women who have lived in the United States or other developed nation for less than 10 consecutive years
* Multiple infants born to one mother
* Plan to feed infants solid foods before infants turn 5 months of age
* Family history of cow milk or soy allergy and/or infants allergic to cow milk protein or soy
* Infants born by C-section
* Infants born with medical complications such as: respiratory distress syndrome, birth defects, and infection
* Infants who have taken antibiotics 4 weeks before enrollment and more than one course of antibiotics since birth
* Infants who have taken probiotics since birth
* Plan to administer probiotics to infants or use of probiotics other than the study supplement by infants for the first two months of the study
* Mothers who have a chronic metabolic disease or obesity
* Mothers who currently smoke or plan to resume smoking during the study period
* Infants who consume solid foods or other liquids other than breastmilk, infant formula or water

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-05-16 (Actual)

PRIMARY OUTCOMES:
Infant fecal B. infantis | Change from baseline to day 280
  The change in infant fecal B. infantis before, during and after supplementation.
Infant fecal Bifidobacterium | Change from baseline to day 280
  The change in infant fecal Bifidobacterium before, during, and after supplementation.
Infant fecal total bacteria | Change from baseline to day 280
  The change in infant fecal total bacteria before, during and after supplementation.
Infant fecal microbiome | Change from baseline to day 280
  The change in infant fecal microbiome before, during and after supplementation.
Infant gastrointestinal symptoms | Change from baseline to day 50
  Gastrointestinal symptoms and related symptoms (discomfort passing bowel movements, vomiting, constipation, colic or irritability) before, during and after supplementation will be determined and reported daily by parental self-report questionnaire.
Infant health status | Change from baseline to day 280
  General health status of the infant such as occurrence of any illness, health care visits for sickness, fever, antibiotic and medication use and parental assessments of infant's overall health.

SECONDARY OUTCOMES:
Maternal secretor status | Change from baseline to day 280
  Determine the relationship between human milk oligosaccharides in breast milk and infant fecal microbiome.
Infant fecal sialic acid concentrations | Change from baseline to day 280
  The change in infant fecal sialic acid and fucose concentrations before, during and after supplementation in infant stool samples.
Infant fecal microbiome and lifestyle | Change from baseline to day 280
  Determine the relationship between the following factors determined by self-report questionnaires: parity, maternal and infant antibiotic intake and maternal use of antimicrobials, infant intake of formula; and the change infant fecal microbiome.
Infant weight | Change from baseline to day 280
  Determine the relationship between infant weight and change in fecal microbiome.
Infant fecal short chain fatty acids | Change from baseline to day 280
  Determine the relationship between fecal short chain fatty acids and fecal microbiome.
Infant gastrointestinal function | Change from baseline to day 280
  Determine the relationship between GI function (fecal inflammatory, GI barrier mediators, LPS) and fecal microbiome.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Smilowitz, PhD, Principal Investigator — University of California, Davis; Mark Underwood, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States

REFERENCES:
- [Background] Bager P, Wohlfahrt J, Westergaard T. Caesarean delivery and risk of atopy and allergic disease: meta-analyses. Clin Exp Allergy. 2008 Apr;38(4):634-42. doi: 10.1111/j.1365-2222.2008.02939.x. Epub 2008 Feb 11. PMID 18266879
- [Background] Thavagnanam S, Fleming J, Bromley A, Shields MD, Cardwell CR. A meta-analysis of the association between Caesarean section and childhood asthma. Clin Exp Allergy. 2008 Apr;38(4):629-33. doi: 10.1111/j.1365-2222.2007.02780.x. PMID 18352976
- [Background] Negele K, Heinrich J, Borte M, von Berg A, Schaaf B, Lehmann I, Wichmann HE, Bolte G; LISA Study Group. Mode of delivery and development of atopic disease during the first 2 years of life. Pediatr Allergy Immunol. 2004 Feb;15(1):48-54. doi: 10.1046/j.0905-6157.2003.00101.x. PMID 14998382
- [Background] Renz-Polster H, David MR, Buist AS, Vollmer WM, O'Connor EA, Frazier EA, Wall MA. Caesarean section delivery and the risk of allergic disorders in childhood. Clin Exp Allergy. 2005 Nov;35(11):1466-72. doi: 10.1111/j.1365-2222.2005.02356.x. PMID 16297144
- [Background] Eggesbo M, Botten G, Stigum H, Nafstad P, Magnus P. Is delivery by cesarean section a risk factor for food allergy? J Allergy Clin Immunol. 2003 Aug;112(2):420-6. doi: 10.1067/mai.2003.1610. PMID 12897751
- [Background] Lewis ZT, Totten SM, Smilowitz JT, Popovic M, Parker E, Lemay DG, Van Tassell ML, Miller MJ, Jin YS, German JB, Lebrilla CB, Mills DA. Maternal fucosyltransferase 2 status affects the gut bifidobacterial communities of breastfed infants. Microbiome. 2015 Apr 10;3:13. doi: 10.1186/s40168-015-0071-z. eCollection 2015. PMID 25922665
- [Background] Ninonuevo MR, Park Y, Yin H, Zhang J, Ward RE, Clowers BH, German JB, Freeman SL, Killeen K, Grimm R, Lebrilla CB. A strategy for annotating the human milk glycome. J Agric Food Chem. 2006 Oct 4;54(20):7471-80. doi: 10.1021/jf0615810. PMID 17002410
- [Background] Ninonuevo MR, Perkins PD, Francis J, Lamotte LM, LoCascio RG, Freeman SL, Mills DA, German JB, Grimm R, Lebrilla CB. Daily variations in oligosaccharides of human milk determined by microfluidic chips and mass spectrometry. J Agric Food Chem. 2008 Jan 23;56(2):618-26. doi: 10.1021/jf071972u. Epub 2007 Dec 19. PMID 18088092
- [Background] Ninonuevo MR, Ward RE, LoCascio RG, German JB, Freeman SL, Barboza M, Mills DA, Lebrilla CB. Methods for the quantitation of human milk oligosaccharides in bacterial fermentation by mass spectrometry. Anal Biochem. 2007 Feb 1;361(1):15-23. doi: 10.1016/j.ab.2006.11.010. Epub 2006 Nov 27. PMID 17181994
- [Background] Sela DA, Chapman J, Adeuya A, Kim JH, Chen F, Whitehead TR, Lapidus A, Rokhsar DS, Lebrilla CB, German JB, Price NP, Richardson PM, Mills DA. The genome sequence of Bifidobacterium longum subsp. infantis reveals adaptations for milk utilization within the infant microbiome. Proc Natl Acad Sci U S A. 2008 Dec 2;105(48):18964-9. doi: 10.1073/pnas.0809584105. Epub 2008 Nov 24. PMID 19033196
- [Background] Sela DA. Bifidobacterial utilization of human milk oligosaccharides. Int J Food Microbiol. 2011 Sep 1;149(1):58-64. doi: 10.1016/j.ijfoodmicro.2011.01.025. Epub 2011 Jan 26. PMID 21342711
- [Background] Sela DA, Garrido D, Lerno L, Wu S, Tan K, Eom HJ, Joachimiak A, Lebrilla CB, Mills DA. Bifidobacterium longum subsp. infantis ATCC 15697 alpha-fucosidases are active on fucosylated human milk oligosaccharides. Appl Environ Microbiol. 2012 Feb;78(3):795-803. doi: 10.1128/AEM.06762-11. Epub 2011 Dec 2. PMID 22138995
- [Background] Sela DA, Li Y, Lerno L, Wu S, Marcobal AM, German JB, Chen X, Lebrilla CB, Mills DA. An infant-associated bacterial commensal utilizes breast milk sialyloligosaccharides. J Biol Chem. 2011 Apr 8;286(14):11909-18. doi: 10.1074/jbc.M110.193359. Epub 2011 Feb 2. PMID 21288901
- [Background] Garrido D, Barile D, Mills DA. A molecular basis for bifidobacterial enrichment in the infant gastrointestinal tract. Adv Nutr. 2012 May 1;3(3):415S-21S. doi: 10.3945/an.111.001586. PMID 22585920
- [Background] Garrido D, Kim JH, German JB, Raybould HE, Mills DA. Oligosaccharide binding proteins from Bifidobacterium longum subsp. infantis reveal a preference for host glycans. PLoS One. 2011 Mar 15;6(3):e17315. doi: 10.1371/journal.pone.0017315. PMID 21423604
- [Background] Garrido D, Nwosu C, Ruiz-Moyano S, Aldredge D, German JB, Lebrilla CB, Mills DA. Endo-beta-N-acetylglucosaminidases from infant gut-associated bifidobacteria release complex N-glycans from human milk glycoproteins. Mol Cell Proteomics. 2012 Sep;11(9):775-85. doi: 10.1074/mcp.M112.018119. Epub 2012 Jun 27. PMID 22745059
- [Background] Garrido D, Ruiz-Moyano S, Jimenez-Espinoza R, Eom HJ, Block DE, Mills DA. Utilization of galactooligosaccharides by Bifidobacterium longum subsp. infantis isolates. Food Microbiol. 2013 Apr;33(2):262-70. doi: 10.1016/j.fm.2012.10.003. Epub 2012 Oct 22. PMID 23200660
- [Background] Garrido D, Ruiz-Moyano S, Mills DA. Release and utilization of N-acetyl-D-glucosamine from human milk oligosaccharides by Bifidobacterium longum subsp. infantis. Anaerobe. 2012 Aug;18(4):430-5. doi: 10.1016/j.anaerobe.2012.04.012. Epub 2012 May 9. PMID 22579845
- [Background] Marcobal A, Barboza M, Froehlich JW, Block DE, German JB, Lebrilla CB, Mills DA. Consumption of human milk oligosaccharides by gut-related microbes. J Agric Food Chem. 2010 May 12;58(9):5334-40. doi: 10.1021/jf9044205. PMID 20394371
- [Background] LoCascio RG, Ninonuevo MR, Freeman SL, Sela DA, Grimm R, Lebrilla CB, Mills DA, German JB. Glycoprofiling of bifidobacterial consumption of human milk oligosaccharides demonstrates strain specific, preferential consumption of small chain glycans secreted in early human lactation. J Agric Food Chem. 2007 Oct 31;55(22):8914-9. doi: 10.1021/jf0710480. Epub 2007 Oct 5. PMID 17915960
- [Background] LoCascio RG, Desai P, Sela DA, Weimer B, Mills DA. Broad conservation of milk utilization genes in Bifidobacterium longum subsp. infantis as revealed by comparative genomic hybridization. Appl Environ Microbiol. 2010 Nov;76(22):7373-81. doi: 10.1128/AEM.00675-10. Epub 2010 Aug 27. PMID 20802066
- [Background] Zivkovic AM, Lewis ZT, German JB, Mills DA. Establishment of a milk-oriented microbiota (MOM) in early life: How babies meet their MOMs. . Functional Food Reviews. 2013;5:3-12.
- [Background] Stark PL, Lee A. The microbial ecology of the large bowel of breast-fed and formula-fed infants during the first year of life. J Med Microbiol. 1982 May;15(2):189-203. doi: 10.1099/00222615-15-2-189. PMID 7143428
- [Background] Haarman M, Knol J. Quantitative real-time PCR assays to identify and quantify fecal Bifidobacterium species in infants receiving a prebiotic infant formula. Appl Environ Microbiol. 2005 May;71(5):2318-24. doi: 10.1128/AEM.71.5.2318-2324.2005. PMID 15870317
- [Background] Penders J, Thijs C, Vink C, Stelma FF, Snijders B, Kummeling I, van den Brandt PA, Stobberingh EE. Factors influencing the composition of the intestinal microbiota in early infancy. Pediatrics. 2006 Aug;118(2):511-21. doi: 10.1542/peds.2005-2824. PMID 16882802
- [Background] Penders J, Gerhold K, Stobberingh EE, Thijs C, Zimmermann K, Lau S, Hamelmann E. Establishment of the intestinal microbiota and its role for atopic dermatitis in early childhood. J Allergy Clin Immunol. 2013 Sep;132(3):601-607.e8. doi: 10.1016/j.jaci.2013.05.043. Epub 2013 Jul 27. PMID 23900058
- [Background] Benno Y, Sawada K, Mitsuoka T. The intestinal microflora of infants: composition of fecal flora in breast-fed and bottle-fed infants. Microbiol Immunol. 1984;28(9):975-86. doi: 10.1111/j.1348-0421.1984.tb00754.x. PMID 6513816
- [Background] Mitsuoka T, Kaneuchi C. Ecology of the bifidobacteria. Am J Clin Nutr. 1977 Nov;30(11):1799-810. doi: 10.1093/ajcn/30.11.1799. No abstract available. PMID 920640
- [Background] Penders J, Vink C, Driessen C, London N, Thijs C, Stobberingh EE. Quantification of Bifidobacterium spp., Escherichia coli and Clostridium difficile in faecal samples of breast-fed and formula-fed infants by real-time PCR. FEMS Microbiol Lett. 2005 Feb 1;243(1):141-7. doi: 10.1016/j.femsle.2004.11.052. PMID 15668012
- [Background] Bezirtzoglou E, Tsiotsias A, Welling GW. Microbiota profile in feces of breast- and formula-fed newborns by using fluorescence in situ hybridization (FISH). Anaerobe. 2011 Dec;17(6):478-82. doi: 10.1016/j.anaerobe.2011.03.009. Epub 2011 Apr 8. PMID 21497661
- [Background] Harmsen HJ, Wildeboer-Veloo AC, Raangs GC, Wagendorp AA, Klijn N, Bindels JG, Welling GW. Analysis of intestinal flora development in breast-fed and formula-fed infants by using molecular identification and detection methods. J Pediatr Gastroenterol Nutr. 2000 Jan;30(1):61-7. doi: 10.1097/00005176-200001000-00019. PMID 10630441
- [Background] Yoshioka H, Iseki K, Fujita K. Development and differences of intestinal flora in the neonatal period in breast-fed and bottle-fed infants. Pediatrics. 1983 Sep;72(3):317-21. PMID 6412205
- [Background] Matsuki T, Watanabe K, Tanaka R, Fukuda M, Oyaizu H. Distribution of bifidobacterial species in human intestinal microflora examined with 16S rRNA-gene-targeted species-specific primers. Appl Environ Microbiol. 1999 Oct;65(10):4506-12. doi: 10.1128/AEM.65.10.4506-4512.1999. PMID 10508082
- [Background] Kleessen B, Bunke H, Tovar K, Noack J, Sawatzki G. Influence of two infant formulas and human milk on the development of the faecal flora in newborn infants. Acta Paediatr. 1995 Dec;84(12):1347-56. doi: 10.1111/j.1651-2227.1995.tb13567.x. PMID 8645949
- [Background] Underwood MA, Kalanetra KM, Bokulich NA, Lewis ZT, Mirmiran M, Tancredi DJ, Mills DA. A comparison of two probiotic strains of bifidobacteria in premature infants. J Pediatr. 2013 Dec;163(6):1585-1591.e9. doi: 10.1016/j.jpeds.2013.07.017. Epub 2013 Aug 29. PMID 23993139
- [Background] Macfarlane GT, Steed H, Macfarlane S. Bacterial metabolism and health-related effects of galacto-oligosaccharides and other prebiotics. J Appl Microbiol. 2008 Feb;104(2):305-44. doi: 10.1111/j.1365-2672.2007.03520.x. PMID 18215222
- [Background] Barile D, Guinard J, Meyrand M, German JB. Examining bioactive components of milk: complex oligosaccharides. AgroFood. 2011;22(4):12-6.
- [Background] Barile D, Marotta M, Chu C, Mehra R, Grimm R, Lebrilla CB, German JB. Neutral and acidic oligosaccharides in Holstein-Friesian colostrum during the first 3 days of lactation measured by high performance liquid chromatography on a microfluidic chip and time-of-flight mass spectrometry. J Dairy Sci. 2010 Sep;93(9):3940-9. doi: 10.3168/jds.2010-3156. PMID 20723667
- [Background] Barile D, Meyrand M, Lebrilla CB, German JB. Examining bioactive components of milk Sources of complex oligosaccharides (Part 2). Agro Food Industry Hi-Tech. 2011;22(4):37-9.
- [Background] Barile D, Rastall RA. Human milk and related oligosaccharides as prebiotics. Curr Opin Biotechnol. 2013 Apr;24(2):214-9. doi: 10.1016/j.copbio.2013.01.008. Epub 2013 Feb 19. PMID 23434179
- [Background] Tao N, DePeters EJ, Freeman S, German JB, Grimm R, Lebrilla CB. Bovine milk glycome. J Dairy Sci. 2008 Oct;91(10):3768-78. doi: 10.3168/jds.2008-1305. PMID 18832198
- [Background] Tao N, DePeters EJ, German JB, Grimm R, Lebrilla CB. Variations in bovine milk oligosaccharides during early and middle lactation stages analyzed by high-performance liquid chromatography-chip/mass spectrometry. J Dairy Sci. 2009 Jul;92(7):2991-3001. doi: 10.3168/jds.2008-1642. PMID 19528576
- [Background] Neville MC, Keller R, Seacat J, Lutes V, Neifert M, Casey C, Allen J, Archer P. Studies in human lactation: milk volumes in lactating women during the onset of lactation and full lactation. Am J Clin Nutr. 1988 Dec;48(6):1375-86. doi: 10.1093/ajcn/48.6.1375. PMID 3202087
- [Background] Dewey KG, Heinig MJ, Nommsen LA, Lonnerdal B. Maternal versus infant factors related to breast milk intake and residual milk volume: the DARLING study. Pediatrics. 1991 Jun;87(6):829-37. PMID 2034486
- [Background] Bekkali N, Hamers SL, Reitsma JB, Van Toledo L, Benninga MA. Infant stool form scale: development and results. J Pediatr. 2009 Apr;154(4):521-526.e1. doi: 10.1016/j.jpeds.2008.10.010. Epub 2008 Dec 3. PMID 19054528
- [Background] Totten SM, Zivkovic AM, Wu S, Ngyuen U, Freeman SL, Ruhaak LR, Darboe MK, German JB, Prentice AM, Lebrilla CB. Comprehensive profiles of human milk oligosaccharides yield highly sensitive and specific markers for determining secretor status in lactating mothers. J Proteome Res. 2012 Dec 7;11(12):6124-33. doi: 10.1021/pr300769g. Epub 2012 Nov 19. PMID 23140396
- [Background] Allen SJ, Jordan S, Storey M, Thornton CA, Gravenor M, Garaiova I, Plummer SF, Wang D, Morgan G. Dietary supplementation with lactobacilli and bifidobacteria is well tolerated and not associated with adverse events during late pregnancy and early infancy. J Nutr. 2010 Mar;140(3):483-8. doi: 10.3945/jn.109.117093. Epub 2010 Jan 20. PMID 20089774
- [Background] Meli F, Puccio G, Cajozzo C, Ricottone GL, Pecquet S, Sprenger N, Steenhout P. Growth and safety evaluation of infant formulae containing oligosaccharides derived from bovine milk: a randomized, double-blind, noninferiority trial. BMC Pediatr. 2014 Dec 20;14:306. doi: 10.1186/s12887-014-0306-3. PMID 25527244
- [Background] Floch MH, Montrose DC. Use of probiotics in humans: an analysis of the literature. Gastroenterol Clin North Am. 2005 Sep;34(3):547-70, x. doi: 10.1016/j.gtc.2005.05.004. No abstract available. PMID 16084313
- [Background] Galdeano CM, de Moreno de LeBlanc A, Vinderola G, Bonet ME, Perdigon G. Proposed model: mechanisms of immunomodulation induced by probiotic bacteria. Clin Vaccine Immunol. 2007 May;14(5):485-92. doi: 10.1128/CVI.00406-06. Epub 2007 Mar 14. No abstract available. PMID 17360855
- [Background] Rosenfeldt V, Benfeldt E, Valerius NH, Paerregaard A, Michaelsen KF. Effect of probiotics on gastrointestinal symptoms and small intestinal permeability in children with atopic dermatitis. J Pediatr. 2004 Nov;145(5):612-6. doi: 10.1016/j.jpeds.2004.06.068. PMID 15520759
- [Background] Klaenhammer TR, Kleerebezem M, Kopp MV, Rescigno M. The impact of probiotics and prebiotics on the immune system. Nat Rev Immunol. 2012 Oct;12(10):728-34. doi: 10.1038/nri3312. PMID 23007572
- [Background] Gratz SW, Mykkanen H, El-Nezami HS. Probiotics and gut health: a special focus on liver diseases. World J Gastroenterol. 2010 Jan 28;16(4):403-10. doi: 10.3748/wjg.v16.i4.403. PMID 20101763
- [Background] Alfaleh K, Anabrees J, Bassler D, Al-Kharfi T. Probiotics for prevention of necrotizing enterocolitis in preterm infants. Cochrane Database Syst Rev. 2011 Mar 16;(3):CD005496. doi: 10.1002/14651858.CD005496.pub3. PMID 21412889
- [Background] Pelucchi C, Chatenoud L, Turati F, Galeone C, Moja L, Bach JF, La Vecchia C. Probiotics supplementation during pregnancy or infancy for the prevention of atopic dermatitis: a meta-analysis. Epidemiology. 2012 May;23(3):402-14. doi: 10.1097/EDE.0b013e31824d5da2. PMID 22441545
- [Background] Degnan FH. The US Food and Drug Administration and probiotics: regulatory categorization. Clin Infect Dis. 2008 Feb 1;46 Suppl 2:S133-6; discussion S144-51. doi: 10.1086/523324. PMID 18181719